CLINICAL TRIAL: NCT01135394
Title: Pharmacogenomics of Thiazolidinediones
Acronym: PPAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Soren Snitker, MD, PhD, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00043497; R01DK074828 (NIH)
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Diabetes
Keywords: Pioglitazone; Type 2 diabetes; Insulin sensitivity; Healthy adults; Thiazolidinediones; Pharmacogenetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pioglitazone (Actos) (Experimental): Participants will have metabolism studies to consist of outpatient X-ray and MR measurements of bone density and body composition, metabolic testing (intravenous glucose tolerance test), and muscle and adipose tissue biopsies. Blood will also be drawn for genetic testing and for microarray studies of leukocytes. Upon completion of the above studies, the participant will begin pioglitazone therapy. Every 4 weeks throughout the drug intervention, glycemic control, lipoprotein profile, and weight will be monitored. After 12 weeks of pioglitazone therapy, the X-ray and MR measurements of body composition, the biopsies, microarray studies for leukocytes and the metabolic tests will be repeated.
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — 30 mg tablet once daily for 4 weeks, then increased to 45 mg once daily for an additional 8 weeks. Total dosage period is 12 weeks.
  Other Names: Actos

SUMMARY:
The purpose of this study is to determine predictors of response to pioglitazone, an anti-diabetic medication. The investigators know from randomized clinical trials that some 30% of patients do not respond to this type of medication. There is presently no way to identify this group of patients leading to unnecessary drug exposure and medication costs.

DETAILED DESCRIPTION:
In phase I, subjects who are eligible based on height and weight and general health information will sign informed consent. In phase II, subjects will be screened to ensure that they fit the inclusion/exclusion criteria, including an oral glucose tolerance test. Other blood tests will be performed to check complete blood count, lipids, liver functions and electrolytes.

Qualifying volunteers will enter phase III, which will consist of outpatient radioimaging and body composition, metabolic testing (intravenous glucose tolerance test), and tissue biopsies. Blood will also be drawn for genetic testing and for microarray studies of leukocytes. Written medication information and instructions for pioglitazone, discharge instructions and satisfaction surveys following the tissue biopsy procedures will be given to subjects during the study. During phase IV, subjects will begin pioglitazone therapy. Every 4 weeks throughout the drug intervention, glycemic control, lipoprotein profile, and weight will be monitored. After 12 weeks of pioglitazone therapy, the X-ray and magnetic resonance (MR) measurements of body composition, the biopsies and the metabolic tests performed during phase III will be repeated (phase V), and blood will be drawn for microarray studies of leukocytes.

Thereafter, subjects will have the option to be enrolled in a 10 week, behavioral weight loss program (phase VI). Following the 10-week weight loss program, a few outcome measurements will be repeated (phase VII).

Throughout the study, Women of Child Bearing Potential (WCBP) will have human human chorionic gonadotrophin (HCG) urine pregnancy tests. Pregnancy tests will only be performed on Women of childbearing potential, meaning women who are pre-menopausal and who have not had surgical sterilization. Women who have not had a hysterectomy or tubal ligation at least six months prior to signing informed consent or have been postmenopausal for at least one year, will be instructed to practice one of the following methods of birth control throughout the study: oral, transdermal, or implantable hormonal contraceptives, intrauterine device, diaphragm plus spermicide, condom plus spermicide, or abstinence. Pioglitazone may reduce the effectiveness of some hormonal types of contraceptives. Women using hormonal methods of birth control will be advised to use a barrier method as well. Female subjects are informed to notify the investigators immediately if they think they might have become pregnant during the study.

Participants who are eligible have 10 visits over an approximate 15-week period. Participants can choose to participate in an optional weight management program for an additional 10 weeks after treatment and before their final visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-64
* BMI: ≥ 25 and ≤ 40

Exclusion Criteria:

* Pregnancy as determined by urine pregnancy test Breast-feeding, or planning to become pregnant during the study
* Physical dimensions exceeding the limits of any equipment used
* Stage III or greater congestive heart failure
* Symptomatic peripheral vascular disease
* Stroke
* Severe hypertension (>170/100 mmHg)
* Anemia (Hgb and Hct < normal reference range)
* Receiving treatment for thyroid, pituitary, kidney or liver disease (except controlled thyroid hormone replacement)
* History of diabetes (as told by doctor, or taking diabetic medications Fasting glucose value diagnostic for diabetes 2-h oral glucose tolerance test diagnostic for diabetes
* Rheumatoid arthritis
* History of wrist, hip or leg fracture after the age of 45
* History of kidney stones
* Medications that the investigator judges will make interpretation of the results difficult or increase the risk of participation (e.g. anticoagulants)
* Any disease or condition that the investigator judges will affect bone metabolism or make interpretation of the results difficult or increase the risk of participation (e.g. anemia, cardiac decompensation, intolerance to pioglitazone, lidocaine, or other agents used)

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2009-03; Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soren Snitker, MD, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was through advertisements in local publications and bulletin boards in the University of Maryland and Baltimore area. Additional recruitment among the Old Order Amish was through the University of Maryland Amish Research Clinic in Lancaster County, Pennsylvania.
Pre-assignment Details: Screening assessments done following informed consent include anthropometry, screening bloodwork, medical history and baseline study assessments. Participants may be excluded prior to start of study drug and/or baseline assessments if they do not meet eligibility criteria.
Groups:
- Pioglitazone (Actos): Participants will have metabolism studies to consist of outpatient X-ray and magnetic resonance (MR) measurements of bone density and body composition, metabolic testing (intravenous glucose tolerance test), and muscle and adipose tissue biopsies. Blood will also be drawn for genetic testing and for microarray studies of leukocytes. Upon completion of the above studies, the participant will begin pioglitazone therapy. Every 4 weeks throughout the drug intervention, glycemic control, lipoprotein profile, and weight will be monitored. After 12 weeks of pioglitazone therapy, the X-ray and MR measurements of body composition, the biopsies, microarray studies for leukocytes and the metabolic tests will be repeated.
  Pioglitazone: 30 mg tablet once daily for 4 weeks, then increased to 45 mg once daily for an additional 8 weeks. Total dosage period is 12 weeks.
Period: Screening
Arm/Group | Pioglitazone (Actos)
Started | 114
Completed | 81
Not Completed | 33
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 10
Not completed — Screening failure | 16
Not completed — Physician Decision | 5
Period: Baseline Assessment
Arm/Group | Pioglitazone (Actos)
Started | 81
Completed | 66
Not Completed | 15
Not completed — Withdrawal by Subject | 9
Not completed — Physician Decision | 3
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 1
Period: Study Treatment
Arm/Group | Pioglitazone (Actos)
Started | 66
Completed | 62
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pioglitazone (Actos)
Number analyzed (Participants) | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 114
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 106
  More than one race | 0
  Unknown or Not Reported | 0
Insulin resistance [Mean (Standard Deviation); unit: HOMA-IR index is unitless by definition] — Homeostatic Model of Insulin Resistance (HOMA-IR) index was calculated as (glucose (mg/dL) x insulin (μU/mL)/405) based on an intravenous glucose tolerance test as per Turner et al.* By definition, HOMA-IR index is unitless.
  *Turner R.C., et al. (1979). "Insulin deficiency and insulin resistance interaction in diabetes: estimation of their relative contribution by feedback analysis from basal plasma insulin and glucose concentrations". Metabolism. 28 (11): 1086-96 Population: HOMA-IR index was calculated only on subjects who had complete data including both intravenous glucose tolerance tests
  HOMA-IR index is unitless by definition
    number analyzed (Participants) | 59
    (all) | 2.74 (1.82)

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Resistance
Description: Change in insulin resistance was calculated as change (end of treatment minus baseline) in HOMA-IR index (glucose (mg/dL) x insulin (μU/mL)/405)
Time Frame: 12 weeks
Population: Included subjects are those who had complete data, including HOMA-IR index at both baseline and after treatment.
Measure: Mean (Standard Deviation); unit: HOMA-IR index is unitless by definition
Groups:
- Pioglitazone (Actos): The study is a one-arm design.
  All participants will receive Pioglitazone: 30 mg tablet once daily for 4 weeks, then increased to 45 mg once daily for an additional 8 weeks. Total dosage period is 12 weeks.
Arm/Group | Pioglitazone (Actos)
Number analyzed (Participants) | 59
HOMA-IR index is unitless by definition | -0.83 (1.23)
Statistical Analysis 1: Comparison: Pioglitazone (Actos); After the change (end-of-treatment minus baseline) in HOMA-IR index had been calculated for each subject, the change (end-of-treatment minus baseline) in expression of each of approximately 45,000 transcripts contained in a human gene array was calculated. A Pearson correlation p-value was calculated for the correlation between change in gene expression and change in HOMA-IR index, with the purpose of identifying the genes whose expression changed in concert with changes in HOMA-IR index; Test type: Other — The genes with p-values below 10^-6 were identified; p < 0.0000001, Genes with p-values below 10^-6 — The genes with p-values below 10^-6 were identified; Pearson correlation p-value = 0.0000001; The genes with P-values below 10^-6 were identified

2. Secondary Outcome: Number of Genes Determined to be Correlated With Change in Insulin Sensitivity
Description: Number of genes determined to be correlated with change in insulin sensitivity as determined by HOMA-IR with a p-value below 0.000001
Time Frame: 12 weeks
Population: Only subjects who had complete RNAseq (RNA sequencing) data and HOMA-IR were included
Measure: Number; unit: Genes
Units Other Than Participants: Genes
Arm/Group | Pioglitazone (Actos)
Number analyzed (Participants) | 55
Number analyzed (Genes) | 53934
Genes | 7

ADVERSE EVENTS:
Time Frame: 12 weeks (treatment phase) + 4 weeks (follow-up) = 16 weeks
Arm/Group | Pioglitazone (Actos)
All-Cause Mortality (participants affected / at risk) | 0/114
Serious Adverse Events (participants affected / at risk) | 2/114
Other Adverse Events (participants affected / at risk) | 15/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (Actos) (N=114)
hypoglycemia (Endocrine disorders) | 1 (2)
Vasovagal response (Cardiac disorders) | 1 (1) — bradycardia secondary to vasovagal response during fat biopsy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (Actos) (N=114)
Hematoma at abdominal fat biopsy site (Skin and subcutaneous tissue disorders) | 7 (7) — Hematoma at abdominal fat biopsy site
Hypoglycemia during intravenous glucose tolerance test (Endocrine disorders) | 8 (9) — Hypoglycemia during intravenous glucose tolerance test

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2006-11-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT01135394/Prot_SAP_000.pdf